CLINICAL TRIAL: NCT02099786
Title: Comprehensive Ototoxicity Monitoring Program for VA: A Randomized Trial
Brief Title: Randomized Trial Comparison of Ototoxicity Monitoring Programs
Acronym: COMP-VA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C0239-R; 3114 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2014-02-26; First posted 2014-03-31 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Cisplatin Ototoxicity; Hearing Loss
Keywords: hearing; cisplatin; Ototoxicity; Veterans
MeSH Terms: conditions — Hearing Loss; Ototoxicity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COMP-VA (Experimental): Hearing testing at each treatment and at 1 month following treatment.
  Interventions: Other: COMP-VA
- Usual Care (Experimental): Hearing testing done according to Audiology Clinic protocol
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: COMP-VA — Hearing testing at each treatment interval by the comp-va audiologist
  Arms: COMP-VA
Other: Standard of care — Hearing testing done in the audiology clinic after oncology referral or patient self referral
  Arms: Usual Care

SUMMARY:
This study involves research. Some chemotherapeutic drugs that can permanently reduce hearing are termed "ototoxic". One such drug is the chemotherapy called cisplatin. Currently, if a patient is receiving cisplatin, hearing is tested in the Audiology Clinic using lengthy protocols and may be retested only when it is requested by their oncologist and when the Veteran can arrange an appointment. Researchers think that hearing testing prior to every treatment of cisplatin may reduce the number of Veterans who get disabling hearing loss from treatment. The purpose of this study is to compare the current method of monitoring hearing (audiology clinic protocols termed "usual care") with a new portable hearing monitoring program (a comprehensive program of ototoxicity monitoring termed "COMP-VA") that tests hearing using a portable hearing testing audiometer and a variety of efficient tools and techniques so that testing can occur prior to each cisplatin treatment at any quiet location in the hospital.

DETAILED DESCRIPTION:
Research objectives are to compare the effectiveness of ototoxicity monitoring implemented using Comp-VA or usual care with regard to (1) improving Veterans' hearing and quality of life outcomes, (2) assisting oncologists in pre-treatment counseling and therapeutic planning and (3) increasing use of post-treatment rehabilitative services.

The investigators plan to recruit a total of 320 Veterans undergoing cisplatin chemotherapeutic treatment over 4 years and 120 control subjects.

Program Evaluation: Hearing testing prior to treatment will be done in order to establish eligibility, enroll and randomize each subject into one of two study arms. At 5 weeks and at one year post-randomization hearing will be re-tested in order to obtain an estimate of longitudinal trends in hearing and quality of life assessment. Use of audiological services following treatment from the randomized subjects will be tracked. Finally, data will also be collected at each treatment interval to track use of counseling tools and oncology personnel treatment decisions.

Serial measurements from subjects receiving cisplatin prior to treatment who are randomized to:

Comp-VA group will get a screening hearing test prior to treatment, at each treatment interval and at one-month post-treatment. Auditory testing will be done on or near the Chemo Unit and will include otoscopy, immittance testing, and a hearing testing done by the Veteran using a self-testing procedure, and may be tested using distortion product otoacoustic emissions (DPOAEs), if they cannot take a reliable hearing test.

Usual care group will receive a full audiometric evaluation (otoscopy, immittance testing, air conduction and bone conduction hearing testing, speech audiometry, and distortion product otoacoustic emissions, DPOAEs) scheduled in the audiology clinic sound booth according to Audiology Service ototoxicity monitoring protocols. Testing will be arranged according to availability of appointments and patient convenience.

Additionally data will also be collected from control subjects who are similar in age and are tested at intervals similar to the chemotherapy subjects.

ELIGIBILITY:
Inclusion Criteria:

All Veterans entering cisplatin chemotherapy will be informed of the project and invited to participate unless the Veteran was excluded by CPRS review or medical advice.

Exclusion Criteria:

* Experimental subjects must be prescribed cisplatin for treatment of cancer to be enrolled in the treatment arms of this study.

Criteria for excluding subjects (chemotherapy and controls subjects) from this study will be:

* cognitively or physically unable to participate (patient or nurse report patient is incapable of participating), CPRS indication that subject exhibits aggressive behavior, subject has documented dementia, Alzheimer's disease, or severe psychosocial disorder, CPRS notes indicate individual is not legally capable of providing informed consent (subject has a legal guardian)
* unable to provide reliable behavioral hearing test responses (for either program evaluation hearing test or baseline, pre -treatment hearing test) as indicated by intra-session behavioral threshold reliability criterion of > +5 dB)
* exhibits Meniere's disease or retrocochlear disorder based on hearing test results, patient report or notes in CPRS
* exhibits active or recent history of middle ear disorder based on otoscopy, tympanometry, patient report, or notes in CPRS
* unwilling to participate
* hearing thresholds > 70 dB SPL at 4 kHz and below (based on DPOAE 'no response' data from a similar protocol described in Bibliography Reference 32, Table 3). The last exclusion was adopted in an effort to increase the potential that DPOAEs will be measurable in a large number of subjects.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn L Konrad-Martin, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brungart D, Schurman J, Konrad-Martin D, Watts K, Buckey J, Clavier O, Jacobs PG, Gordon S, Dille MF. Using tablet-based technology to deliver time-efficient ototoxicity monitoring. Int J Audiol. 2018 Sep;57(sup4):S25-S33. doi: 10.1080/14992027.2017.1370138. Epub 2017 Sep 12. PMID 28893111
- [Background] Dille MF, McMillan GP, Helt WJ, Konrad-Martin D, Jacobs P. A Store-and-Forward Tele-Audiology Solution to Promote Efficient Screenings for Ototoxicity during Cisplatin Cancer Treatment. J Am Acad Audiol. 2015 Oct;26(9):750-60. doi: 10.3766/jaaa.15028. PMID 26415968
- [Background] Reavis KM, McMillan GP, Dille MF, Konrad-Martin D. Meta-Analysis of Distortion Product Otoacoustic Emission Retest Variability for Serial Monitoring of Cochlear Function in Adults. Ear Hear. 2015 Sep-Oct;36(5):e251-60. doi: 10.1097/AUD.0000000000000176. PMID 25985018
- [Background] Konrad-Martin D, Knight K, McMillan GP, Dreisbach LE, Nelson E, Dille M. Long-Term Variability of Distortion-Product Otoacoustic Emissions in Infants and Children and Its Relation to Pediatric Ototoxicity Monitoring. Ear Hear. 2020 Mar/Apr;41(2):239-253. doi: 10.1097/AUD.0000000000000536. PMID 29280917
- [Background] Konrad-Martin D, Poling GL, Garinis AC, Ortiz CE, Hopper J, O'Connell Bennett K, Dille MF. Applying U.S. national guidelines for ototoxicity monitoring in adult patients: perspectives on patient populations, service gaps, barriers and solutions. Int J Audiol. 2018 Sep;57(sup4):S3-S18. doi: 10.1080/14992027.2017.1398421. Epub 2017 Nov 20. PMID 29157038
- [Background] Garinis AC, Cornell A, Allada G, Fennelly KP, Maggiore RJ, Konrad-Martin D. Ototoxicity monitoring through the eyes of the treating physician: Perspectives from pulmonology and medical oncology. Int J Audiol. 2018 Sep;57(sup4):S19-S24. doi: 10.1080/14992027.2017.1381769. Epub 2017 Oct 5. PMID 28978238
- [Background] Konrad-Martin D, Poling GL, Dreisbach LE, Reavis KM, McMillan GP, Lapsley Miller JA, Marshall L. Serial Monitoring of Otoacoustic Emissions in Clinical Trials. Otol Neurotol. 2016 Sep;37(8):e286-94. doi: 10.1097/MAO.0000000000001134. PMID 27518137
- [Background] Konrad-Martin D, Reavis KM, McMillan G, Helt WJ, Dille M. Proposed comprehensive ototoxicity monitoring program for VA healthcare (COMP-VA). J Rehabil Res Dev. 2014;51(1):81-100. doi: 10.1682/JRRD.2013.04.0092. PMID 24805896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-seven Veterans receiving cisplatin for the treatment of cancer were randomized to one of the two treatment arms of the clinical trial. Thirty-six healthy participants were studied to assess normal variability in auditory function measures over time; they were not part of the clinical trial portion of this research project.
Groups:
- Usual Care: Hearing testing done according to Audiology Clinic protocol
  Standard of care: Hearing testing done in the audiology clinic after oncology referral
Period: Overall Study
Arm/Group | COMP-VA | Usual Care
Started | 24 | 23
Program Eval 1 | 24 (Baseline (prior to randomization and first cisplatin dose)) | 23 (Baseline (prior to randomization and first cisplatin dose))
Program Eval 2 | 23 (One month post randomization) | 19 (One month post randomization)
Program Eval 3 | 21 (One year post randomization) | 15 (One year post randomization)
Completed | 21 | 15
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COMP-VA | Usual Care | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (6.4) | 64.7 (9.1) | 64.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 23 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
3, 4, and 6 kHz pure tone average (PTA) [Mean (Standard Deviation); unit: dB HL] | 47.8 (21.5) | 55.4 (19.8) | 51.6 (20.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Ototoxic Hearing Shift
Description: Veterans randomized to the COMP-VA arm will have improved hearing outcomes (a) fewer ASHA-significant threshold shifts, (b) fewer CTCAE grade 1 or greater hearing shifts at Program Evaluation 3 as compared with Veterans randomized to the Usual Care arm.
  1. ASHA Shift is defined as:
     20 dB shift at a single frequency 10 dB shift at two adjacent frequencies loss of response at three adjacent frequencies
  2. CTCAE Grade 1 or greater ototoxicity = hearing shift of 15-25 dB averaged at 2 contiguous test frequencies
Time Frame: 35 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | COMP-VA | Usual Care
Number analyzed (Participants) | 21 | 15
Participants | 15 | 8
Statistical Analysis 1: Comparison: COMP-VA vs Usual Care; Null hypothesis: There is no difference in the number of participants with ASHA-significant threshold shifts between treatment arms; Test type: Superiority; p = .27, Regression, Logistic; Odds Ratio (OR) = 2.2, 95% CI 2-sided [.55 to 8.8]
Statistical Analysis 2: Comparison: COMP-VA vs Usual Care; Null hypothesis: There is no difference in the number of participants with CTCAE grade 1 or greater hearing loss between treatment arms; Test type: Superiority; p = .67, Regression, Logistic; Odds Ratio (OR) = 1.4, 95% CI 2-sided [.3 to 5.9]

2. Primary Outcome: Number of Participants Who Accessed the Audiology Clinic for Aural Rehabilitation
Description: Veterans randomized to Comp-VA will access and use audiology rehabilitation at higher rates than usual care up to 1 year post-treatment. This includes: New hearing aid issued; Hearing aid adjustments made; Technology updated.
Time Frame: through study completion, an average of 1 year post randomization
Population: All participants who received at least one dose of cisplatin and had at least two Program Evaluations.
Measure: Count of Participants; unit: Participants
Arm/Group | COMP-VA | Usual Care
Number analyzed (Participants) | 24 | 23
Participants | 12 | 12
Statistical Analysis 1: Comparison: COMP-VA vs Usual Care; Null hypothesis is no difference in audiology clinic use between treatment arms; Test type: Superiority; p = .88, Regression, Logistic; Odds Ratio (OR) = .92, 95% CI 2-sided [.29 to 2.9]

3. Primary Outcome: Number of Participants With Mortality
Description: Mortality among participants defined as differences in rates of death within one year of randomization.
Time Frame: 1 year post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | COMP-VA | Usual Care
Number analyzed (Participants) | 24 | 23
Participants | 2 | 4
Statistical Analysis 1: Comparison: COMP-VA vs Usual Care; Test type: Non-Inferiority — We require a non-inferiority margin of no more than 1.1 mortality odds among COMP-VA patients relative to Usual Care patients. This means that the upper 95% confidence bound for the fitted odds ratio must be less than 1.1 to reject the null hypothesis that COMP-VA induces extra mortality risk; Odds Ratio (OR) = 1.9

4. Primary Outcome: Hearing-related Quality of Life Measure
Description: Differences in the Hearing Handicap Inventory for Adults (HHIA) questionnaire score [or Hearing Handicap Inventory for the Elderly (HHIE) score as appropriate] depending on the age of the subject.
  Minimum possible value = 0 Maximum possible value = 100 A higher score indicates poorer performance
Time Frame: 1 year post randomization
Population: Missing data on some participants due to loss of follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COMP-VA | Usual Care
Number analyzed (Participants) | 21 | 15
score on a scale | 20.8 (18.6) | 23.2 (22.5)
Statistical Analysis 1: Comparison: COMP-VA vs Usual Care; Test type: Superiority; p = .72, t-test, 2 sided — The a priori threshold for statistical significance is .05

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | COMP-VA | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/24 | 4/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/24 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT02099786/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT02099786/SAP_001.pdf